CLINICAL TRIAL: NCT03113045
Title: Seated Time for Hypotension in Cesarean Delivery: A Biased Coin Design Trial for 90% Efficacy
Brief Title: Seated Time for 90% Incidence of Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Albert Moore, Principle Investigator, Royal Victoria Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15010MUHC
Record Dates: First submitted 2017-03-18; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Masking Description: The observer will not be made aware of the time that the patient will sit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seated Time (Experimental): Pts will be seated for the allocated time depending on the previous patients hypotensive response
  Interventions: Other: seated time

INTERVENTIONS:
Other: seated time — Pt will be seated for a predetermined time period. All Patients will receive intrathecal bupivacaine and morphine.

SUMMARY:
The study will determine the 90% effective seated time after intrathecal injection of hyperbaric bupivacaine to avoid hypotension in patients undergoing cesarean delivery.

DETAILED DESCRIPTION:
The study will use a Biased Coin Design (BCD), up-and-down sequential method, to determine the ET90 for absence of hypotension during Cesarean delivery. In this methodology, the first patient will be assigned an a priori initial seated time. Any other patient will be assigned a seated time based on the presence or absence of hypotension in the previous patient. If the previous patient developed hypotension, then the new patient will be seated for a longer time, which will be equal to the seated time of the previous patient plus a pre-determined time increment (up to an also pre-determined maximum allowed time). If no hypotension occurred to the previous patient, the new patient will be assigned one seated time from two choices: The same seated time that has been assigned to the previous patient, or a seated time shorter than that of the previous patient by a pre-determined time decrement (the pre-determined time increment and decrement are the same). The choice will be determined from a biased coin result, with a probability of 0.9 for assigning 'the same as previous' seated time and a probability of 0.1 for assigning a 'shorter seated time'.

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton pregnancies scheduled for elective cesarean delivery

Exclusion Criteria:

* BMI>35
* Unable to communicate in study language
* ASA greater than 2
* Hypertensive disease of pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Hypotension | 30 minutes
  Presence of hypotension before delivery

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moore, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No